CLINICAL TRIAL: NCT00412165
Title: PACE-iDP: An Intervention for Youth at Risk for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R18DK064321 (NIH); UCSD#: 2006-4039
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Overweight; Diabetes
Keywords: Prevention of Type 2 Diabetes; Adolescents; Obesity; Overweight; Internet Technology; Cell Phone
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus | interventions — Population Groups

ARMS (4):
- usual care (No Intervention): Usual care arm receives standard physical activity, nutrition and weight loss information from their primary care provider. The study offers and pays for a series of weight management sessions provided by Rady's Children's Hospital and Health Center's Nutrition Dept.
- Intervention - Web (Experimental): This group receives access to a program internet site with weekly challenges aimed at weight loss through increased physical activity and nutrition.
  Interventions: Behavioral: Weekly access to interactive web site
- Intervention - Group (Experimental): This group receives access to a program internet site with weekly challenges aimed at weight loss through increased physical activity and nutrition and has access to monthly group session with other teen and parent participants.
  Interventions: Behavioral: Group
- Intervention - Cell Phone (Experimental): This group receives access to a program internet site with weekly challenges aimed at weight loss through increased physical activity and nutrition and are provided with cell phones to use during the program. The cell phone allows for the transfer of text messages from the study to the participant that are tailored to their health goals. In addition, self-monitoring and uploading capabilities to the program website are included.
  Interventions: Behavioral: Cell Phone

INTERVENTIONS:
Behavioral: Cell Phone — The cell phone arm receives access to the website with weekly health ed materials and weekly case management via phone, mail, e-mail
  Arms: Intervention - Cell Phone
Behavioral: Weekly access to interactive web site — This group receives access to the website with weekly health ed materials and weekly case management via phone, mail, e-mail
  Arms: Intervention - Web
Behavioral: Group — The Group arm receives monthly face to face group sessions plus access to the website with weekly health ed materials and weekly case management via phone, mail, e-mail
  Arms: Intervention - Group

SUMMARY:
This randomized control study (sponsored by the NIH, NIDDK) is aimed at reducing BMI in overweight adolescents at risk for the development of type 2 diabetes. The study will examine whether an integrated primary care, web and cell-phone-based intervention can produce initial and sustained improvements in anthropometric, behavioral, metabolic, and physiological outcomes in overweight adolescents. The primary goal is to reduce BMI (Body Mass Index)in overweight adolescents.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (DM) is a common disease that plagues over 16 million adults in the United States (American Diabetes Association [ADA], 2002). Over the past decade, the number of adults diagnosed with diabetes has risen dramatically. The high rates of type 2 diabetes have been associated with the simultaneously rapid increase in the prevalence of obesity, and diminished levels of physical activity in the population (Wing, 2001).

Type 2 diabetes is increasing in children and adolescents in the U.S. and worldwide (ADA, 2000). Several studies have demonstrated higher risk of type 2 diabetes in African-American, Hispanic, and American Indian children and adolescents (Glaser, 1997; Dean, 1992; Pinhas-Hamiel, 1996; Rosenbloom, 1999). Other characteristics, or risk factors, that may be used to identify children at high-risk for developing type 2 diabetes include obesity, family history, and physiologic manifestations of insulin resistance (ADA, 2000). Up to 85% of children with type 2 diabetes are overweight or obese at diagnosis. A majority of children with type 2 diabetes have at least one parent or first-degree relative with type 2 diabetes. Physiologic findings of insulin resistance that are present in large percentages of children with type 2 diabetes include acanthosis nigricans, polycystic ovarian syndrome, hypertension and lipid disorders (ADA, 2000). Among US children, the mean age at diagnosis of type 2 diabetes is between 12 and 14 years (Moran, 1999; Goran MI, 2001).

Obesity is commonly found in children with type 2 diabetes, and the increasing incidence of children with type 2 diabetes has been attributed to the growing problem of pediatric overweight and obesity (Fagot-Camapagna, et.al, 2000). It is often hypothesized that an industrialized, or "Westernized" lifestyle of excessive energy intake and sedentary behavior partially explains the recent emergence of type 2 diabetes and obesity in youth (Hill & Peters, 1998; Koplan & Dietz, 2000). Evidence that the number of years being obese is positively correlated with diabetes risk (Everhart, 1992), supports intervening in adolescence to minimize the number of years of obesity.

Obesity and physical inactivity are thought to be the main modifiable determinants of this disease, and interventions targeting diet and physical activity have been surprisingly effective in preventing diabetes in high-risk adults (Tuomilehto, 2001; NIDDK, 2001). There are no published studies that examine the efficacy of similar lifestyle interventions aimed at children and adolescents. Our rationale for intervening on these behaviors with high-risk adolescents is based on these findings, as well as the following: (a) the majority of adolescents do not meet current guidelines for physical activity and nutrition and (b) there is a steep age-related decline in physical activity that peaks in the teen years. In its March 2000 Consensus Statement of Type 2 Diabetes In Children and Adolescents, the ADA expert panel stated that, "Primary care providers have an obligation to encourage lifestyle modifications that might delay or prevent the onset of type 2 diabetes in children at high risk. Lifestyle interventions focusing on weight management and increasing physical activity should be promoted in all children at high risk for the development of type 2 diabetes." (ADA, 2000).

ELIGIBILITY:
Inclusion Criteria:

Criteria for participation in the study include:

* Being overweight (BMI > 85th percentile for age and sex, weight for height >85th percentile, or weight >120% of ideal for height). In addition, at least half of the study participants will have a BMI > 95th percentile for age and sex. Study participants will have a maximum body weight of 285 pounds.
* Adolescent subjects must also have at least two of the following risk factors:

  * family history of type 2 diabetes in a first-or second-degree relative,
  * race/ethnicity of American Indian, African-American, Hispanic, Asian/Pacific Islander, or
  * signs of insulin resistance (acanthosis nigricans, hypertension, dyslipidemia, or polycystic ovarian syndrome).
* In addition, adolescent subjects must be able to read and speak English or Spanish, have access to the Internet at home, school, or work, be reachable at a telephone number, be willing to participate in monthly 90-minute group meetings, have plans to stay in the San Diego area for the one-year study period, and have an English or Spanish speaking parent/guardian also willing to participate in the study.
* Parental consent (obtained in parents primary language) and subject assent is also required.
* Participants must have a parent or guardian agree to enroll who is able to speak and read in English or Spanish, has ongoing access and uses the internet, and plans to reside in San Diego for the length of the study.

Exclusion Criteria:

Subjects will be excluded from participation if they have any of the following conditions:

* Diabetes
* Pregnancy
* Cardiovascular problem, musculoskeletal problem or any medical condition that would limit their ability to comply with physical activity or dietary recommendations.
* Patients in foster care will be ineligible due to difficulty in obtaining follow-up measures.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect, at 12 months, of the 3 intensities of the PACEi-DP intervention on Body Mass Index (BMI) among male & female adolescents. | baseline, 6 mo, 12 mo

SECONDARY OUTCOMES:
at 6 and 12 months,the impact of the PACEi-DP interventions on:metabolic and physiological manifestations of insulin resistance | 6 mo, 12 mo
anthropometric measures including BMI at 6 months, waist to hip ratio at 6 and 12 months, percent body fat (DEXA) at 6 and 12 months,and | 6 mo, 12 mo
behavioral measures of diet and physical activity. | 6 mo, 12 mo

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD - CALIT2- Atkinson Hall, La Jolla, California, United States

REFERENCES:
- [Derived] Kolodziejczyk JK, Gutzmer K, Wright SM, Arredondo EM, Hill L, Patrick K, Huang JS, Gottschalk M, Norman GJ. Influence of specific individual and environmental variables on the relationship between body mass index and health-related quality of life in overweight and obese adolescents. Qual Life Res. 2015 Jan;24(1):251-61. doi: 10.1007/s11136-014-0745-1. Epub 2014 Jul 1. PMID 24980678
- [Derived] Patrick K, Norman GJ, Davila EP, Calfas KJ, Raab F, Gottschalk M, Sallis JF, Godbole S, Covin JR. Outcomes of a 12-month technology-based intervention to promote weight loss in adolescents at risk for type 2 diabetes. J Diabetes Sci Technol. 2013 May 1;7(3):759-70. doi: 10.1177/193229681300700322. PMID 23759410
- [Derived] Huang JS, Gottschalk M, Norman GJ, Calfas KJ, Sallis JF, Patrick K. Compliance with behavioral guidelines for diet, physical activity and sedentary behaviors is related to insulin resistance among overweight and obese youth. BMC Res Notes. 2011 Feb 1;4:29. doi: 10.1186/1756-0500-4-29. PMID 21281521